CLINICAL TRIAL: NCT03132844
Title: Epidemiological Study on the Vaccination Coverage of the Population Aged 75 Years and Over in Picardy. According to the Study of 200 Patients Followed by General Practitioners of the Somme in 2016.
Acronym: PICARVAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-38 Dr Deschasse
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Vaccination; Elderly
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis records of patients over 75 years of age — Demonstrate the percentage of patients over 75 years of age attending general medicine in the Somme, with an up-to-date vaccination schedule, in view of the HAS 2016 recommendations, for the following vaccines: DTp, influenza, pneumococcus, shingles.

SUMMARY:
In France, the vaccination coverage of seniors is clearly deficient. It seems to be a cultural specificity, dating back more than 100 years, and which does not exist in Scandinavia, nor in much of the Anglo-Saxon world. Only influenza vaccination is a success for seniors. The high public health council sets the objective of immunization coverage in patients over 65 years of age to 80% whether or not the patient is benefiting from an exonerative ALD. The data collections carried out with the various pension funds objective have a lower immunization coverage with a rate ranging from 48.8 to 64%. Thus any medical consultation should be an opportunity to update the vaccination schedule of adults and the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman,> 75 years old.
* Seen in consultation at the doctor's office
* In 2016.

Exclusion Criteria:

* Patient seen during a home visit.
* Patient resident in EHPAD.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 75 years of general practice in the Somme
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Analysis of the rate of patients over 75 years old followed in general medicine in the Somme, with an up-to-date immunization schedule | 5 months
  Analysis of the rate of patients over 75 years old followed in general medicine in the Somme, with an up-to-date immunization schedule

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France